CLINICAL TRIAL: NCT03087968
Title: Evaluation of HepQuant SHUNT to Assess Liver Disease; Substudy Within GS-US-416-2124
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No longer a sub-study - Changing to an independent parallel study
Sponsor: HepQuant, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: HepQuant-002-2124
Record Dates: First submitted 2017-03-09; First posted 2017-03-23 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2017-09

CONDITIONS: Severe Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- GS-4997 + Prednisolone (Experimental): GS-4997 + Prednisolone for 28 days
  HepQuant SHUNT Test
  Interventions: Drug: GS-4997; Drug: Prednisolone; Device: HepQuant SHUNT Test
- Prednisolone + Placebo (Placebo Comparator): Placebo + Prednisolone for 28 days
  HepQuant SHUNT Test
  Interventions: Drug: Prednisolone; Device: HepQuant SHUNT Test; Drug: Placebo

INTERVENTIONS:
Drug: GS-4997 — Experimental drug
  Arms: GS-4997 + Prednisolone
Drug: Prednisolone — Control drug that is also administered with the Experimental drug, GS-4997. This drug is used in both arms.
Device: HepQuant SHUNT Test — The HepQuant SHUNT Liver Diagnostic Kit is intended for use in the quantitative detection of 13C-cholate and d4-cholate in blood serum, collected after the intravenous administration of 13C-cholate and the oral ingestion of d4-cholate. The device is indicated to assess the severity of liver disease.
  For use by health care professionals. Administer the test under a physician's supervision. The HepQuant Analytical Testing Laboratory must analyze the serum samples.
  Other Names: SHUNT
Drug: Placebo — Placebo
  Arms: Prednisolone + Placebo

SUMMARY:
This clinical investigation is a substudy within GS-US-416-2124, IND 129570, which is A Phase 2, Double-Blind, Randomized Study Evaluating the Safety, Tolerability, and Efficacy of GS-4997 in Combination with Prednisolone versus Prednisolone Alone in Subjects with Severe Alcoholic Hepatitis. The use of the HepQuant SHUNT test is to assess liver disease severity before, during, and after treatment with GS-4997 or placebo, to assess liver disease severity.

DETAILED DESCRIPTION:
The main study is a Phase 2, double blind, proof-of-concept, randomized study evaluating the safety, tolerability, and biological activity of GS-4997 in combination with prednisolone, compared to prednisolone alone, in subjects with severe, histologically-confirmed AH.

This substudy uses the HepQuant SHUNT Liver Diagnostic test to assess severity of disease at baseline and to track disease progression or improvement over the 24 weeks of the study. The HepQuant SHUNT test will be performed at baseline (Day 1) and at Weeks 1, 2, 4, 12, and 24 regardless of treatment Arm.

GS-4997 Dose and Mode of Administration. Subjects will be randomized 1:1 to either:

* Treatment Group A: GS-4997 18 mg (1 x 18 mg tablet) AND prednisolone 40 mg (4 x 10 mg tablets), both administered orally once daily
* Treatment Group B: GS-4997 placebo (1 tablet) AND prednisolone 40 mg (4 x 10 mg tablets), both administered orally once daily

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give informed consent prior to any study specific procedures being performed. In individuals with hepatic encephalopathy (HE) which may impair decision-making, consent will be obtained per hospital procedures (eg, by Legally Authorized Representative)
2. Clinical diagnosis of severe AH
3. Maddrey's DF ≥ 32 at screening

Exclusion Criteria:

Key Exclusion Criteria:

1. Pregnant or lactating females;
2. Other causes of liver disease including chronic hepatitis B (hepatitis B surface antigen [HBsAg] positive), chronic hepatitis C (HCV RNA positive), acetaminophen hepatotoxicity, biliary obstruction, and autoimmune liver disease;
3. Serum AST >400 U/L or ALT >300 U/L;
4. MELD >30 at screening;
5. Maddrey's DF >60 at screening;
6. Grade 4 Hepatic Encephalopathy (HE) by West Haven criteria;
7. Concomitant or previous history of hepatocellular carcinoma;
8. History of liver transplantation;
9. HIV Ab positive;
10. Clinical suspicion of pneumonia;
11. Uncontrolled sepsis;
12. Uncontrolled gastrointestinal (GI) bleeding or controlled GI bleeding within 7 days of screening that was associated with shock or required transfusion of more than 3 units of blood;
13. Type 1 hepatorenal syndrome (HRS) or renal failure defined as a serum creatinine >221 μmol/L (>2.5 mg/dL) or the requirement for renal replacement therapy;
14. Individuals dependent on inotropic (eg, epinephrine or norepinephrine) or ventilatory support (ie, endotracheal intubation or positive-pressure ventilation);
15. Portal vein thrombosis;
16. Acute pancreatitis;
17. Cessation of alcohol consumption for more than 2 months before Baseline/ Day 1 NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07-31 (Estimated); Primary Completion 2017-09-13 (Actual); Study Completion 2017-09-13 (Actual)

PRIMARY OUTCOMES:
To compare the change in (DSI ) Disease Severity Index between GS-4997 treatment and placebo arms | HepQuant Shunt testing will be done at baseline (Day1), Week 1, Week 4, Week 12, Week 24
  Using the SHUNT DSI to evaluate the liver, this outcome will compare the two arms to determine if SHUNT DSI is able to measure a change between the experimental and control groups.

SECONDARY OUTCOMES:
Secondary Outcome 1 | HepQuant Shunt testing will be done at baseline (Day1), Week 1, Week 4, Week 12, Week 24
  To determine the relationship of baseline Disease Severity Index (DSI) to mortality risk;
Secondary Outcome 2 | HepQuant Shunt testing will be done at baseline (Day1), Week 1, Week 4, Week 12, Week 24
  To determine the relationship of change in Disease Severity Index (DSI) to mortality risk
Secondary Outcome 3 | HepQuant Shunt testing will be done at baseline (Day1), Week 1, Week 4, Week 12, Week 24
  To correlate baseline Disease Severity Index (DSI) with baseline Maddrey, MELD, and Lille scorestest with the pharmacokinetics of GS-4997
Secondary Outcome 4 | HepQuant Shunt testing will be done at baseline (Day1), Week 1, Week 4, Week 12, Week 24
  To determine the relationship between baseline Disease Severity Index (DSI), Maddrey, MELD, and Lille scores and mortality

CONTACTS AND LOCATIONS:
Overall Officials: Greg Everson, MD, Principal Investigator — HepQuant, LLC
Locations (13):
- United States (13):
  - Southern California Research Center, Coronado, California
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - Liver Institute of Virginia, Newport News, Virginia
  - Liver Institute of Virginia, Richmond, Virginia
  - VCU Health System, Richmond, Virginia
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided